CLINICAL TRIAL: NCT04295291
Title: Quality of Cardiopulmonary Resuscitation Pre- and Intra Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Ostfold University College (Other)
Responsible Party: Principal Investigator, Ann-Chatrin Leonardsen, Associate Professor, Ostfold University College
Other Study IDs: AB 3418
Record Dates: First submitted 2020-01-05; First posted 2020-03-04 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Death; Cardiac Arrest; Cardiac Arrhythmia; Cardiac Disease
Keywords: Cardiopulmonary resuscitation; Defibrillation; Ventilation; Quality; Mortality; Morbidity
MeSH Terms: conditions — Death; Heart Arrest; Arrhythmias, Cardiac; Heart Diseases; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The survival after intrahospital cardiac arrest has been reported to 15%. In Norway this varies between 16 and 23%.). Many factors are associated with survival after cardiac arrest, both intra- and prehospital. Recent studies have not included information about individual patient factors and the outcome after cardiopulmonary resuscitation (CPR). In the current hospital, we are able to record patient specific information related to a cardiac arrest/CPR situation, and thereby be able to assess patient-related factors associated with both detection, treatment and outcome of CPR.

DETAILED DESCRIPTION:
Several factors have been associated with survival, e.g. to monitor hands-off time(Odds ratio, OR, for 2.48, 95% KI 1.11-5.56, p=.03), monthly assessment of all cardiac arrest cases (OR 6.9, 95% KI 1.41-33.92), and includin av local coordinator for CPR (OR 2.93, 95% KI 1.08-7.94, p=.03), as well as depth of compressions. Nevertheless, information about cardiac arrests and CPR have not been assessed in relation to patient specific information. In the current hospital, we are able to record the CPR sequence, and see this in relation to other patient- and case- specific information such as initial cardiac rythm, time to first compression, hands-off time, quality of CPR, and factors affecting the treatment and outcome.

The hospital has 71 registered defibrillators used in CPR. The current study will both gather retrospective data- not seen in relation to patient specific information, and prospective data related to specific patients.

ELIGIBILITY:
Inclusion Criteria:

* cardiac arrest (all reasons)
* a defibrillator has been used
* over 18 years
* cardiopulmonary resuscitation has been conducted

Exclusion Criteria: N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with cardiac arrest, treated with cardio-pumonary resusciation and the use of a defirbillator with USB memory stick installed (all 71 in the current hospital)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | up to 30 days
  Patient dead or alive